CLINICAL TRIAL: NCT00885235
Title: Evaluation of the PillCam Colon Capsule Endoscopy Preparation and Procedure
Brief Title: Evaluation of the PillCam™ Colon Capsule Endoscopy (PCCE) Preparation and Procedure
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MA-101
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2009-08

CONDITIONS: Bowel Diseases
Keywords: Bowel Diseases
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Subjects that are indicated for colonoscopy who are suspected or known to suffer from large bowel diseases.

SUMMARY:
The purpose of this study is to evaluate the effect of the PCCE preparation and procedure on colon cleansing level and excretion rate.

DETAILED DESCRIPTION:
The evaluation of subjects with suspected colonic disease includes endoscopic imaging by colonoscopy and radiologic imaging such as air-contrast barium enema, or CT colonography. The PillCam® platform offers an alternative approach for endoscopic visualization of the colon using capsule endoscopy, an ingestible device which contains imagers, light sources, a power source and a radio frequency transmitter. Advantages of the PillCam® platform include the elimination of the need for sedation, the minimally invasive, painless nature of the exam, and the ability to pursue normal daily activities immediately following the procedure . Furthermore, compared to standard colonoscopy, the PillCam® platform may be more readily accepted by patients and thereby improving compliance with colorectal cancer screening recommendations.

The PillCam® SB capsule (formerly M2A® Capsule) that was cleared by the FDA in August 2001 for small bowel evaluation has been ingested to date by more than 700,000 people worldwide and is well accepted by patients and physicians as well as the major gastrointestinal professional organizations. However, adequate visualization of the colon cannot be achieved with the standard PillCam®SB capsule because of the anatomical and physiological properties of the colon which are significantly different than the small bowel. Moreover, other issues that limit the evaluation of the colonic mucosa by the standard PillCam® SB procedure include an unsatisfactory level of colon cleanliness and slow progression of the PillCam® SB capsule through the colon during the desired examination time. Therefore, the development and introduction of a specially designed, customized colon capsule combined with a specifically designed capsule colonoscopy procedure allows for more efficient evaluation of the colonic mucosa. This is expected to improve the capability of the PillCam® platform to detect colonic pathologies and to serve as a diagnostic and screening tool for colonic disease. Further details of the PillCam™ Colon Capsule Endoscope (PCCE) can be found in the device description section.

This is a pilot study that is designed to develop the optimal PCCE procedure by measuring the levels of cleanliness and capsule excretion rates. Furthermore, capsule endoscopy and colonoscopy procedures will be compared in regards to the detection of polyps and lesions in the colon.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over ≥ 50 years of age scheduled for colorectal cancer screening
* Subjects over ≥ 50 years of age with one or more of the following clinical symptoms: rectal bleeding, hematochezia, melena, positive FOBT, recent change of bowel habits, or diarrhea/constipation of recent onset.
* Subject ≥ 18 years of age with one of the following:

  * Positive findings (≥ 10 mm polyps) in the colon on a GI radiographic study (BE, CT scan, etc) OR
  * Personal history of colorectal cancer (CRC) or adenomatous polyps and ≥5 years since last colonoscopy

Exclusion Criteria:

* Subject has dysphagia or any swallowing disorder
* Subject has congestive heart failure
* Patient has significant renal insufficiency, heart disease or any other condition that the investigator would expect to increase the risk of complications from magnesium citrate, such as dehydration or electrolyte imbalance
* Subject has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator
* Subject has a cardiac pacemaker or other implanted electro medical device.
* Subject has any allergy or other known contraindication to the medications used in the study
* Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Subject with any condition believed to have an increased risk for capsule retention such as Crohn's disease, intestinal tumors, radiation enteritis, or NSAID enteropathy,
* Subject with gastrointestinal motility disorders
* Subject has known delayed gastric emptying
* Subject has any condition, which precludes compliance with study and/or device instructions.
* Women who are either pregnant or nursing at the time of screening, or are of child-bearing potential and do not practice medically acceptable methods of contraception such as: surgical sterilization, approved hormonal contraceptives (i.e. birth control pills, Depo-Provera), barrier methods (i.e. condom or diaphragm) used with a spermicide and an intrauterine device (IUD)
* Subject suffers from life threatening conditions
* Subject currently participating in another clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects that are indicated for colonoscopy who are suspected or known to suffer from large bowel diseases.
  The study population will consist of subjects who fulfill at least one of the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Colon cleansing level score for PCCE | Within 7 days
Grading of visual interference from bubbles in the colon for PCCE | Within 7 days
Number of colon capsules excreted over time | Within 7 Days
Capsule transit time from ingestion to entrance into the cecum & through the colon | Within 7 Days
Number, type and severity of adverse events | WithIn 7 days

SECONDARY OUTCOMES:
Accuracy parameters (sensitivity, specificity ,NPV,PPV,LR) of PCCE in detecting polyps equal to or larger than 10mm as compared to colonoscopy | within 7 days
Accuracy parameters (sensitivity, specificity ,NPV,PPV,LR) of PCCE in detecting polyps equal to or larger than 6mm as compared to colonoscopy | within 7 days
The diagnostic yield of PCCE in detecting a variety of colonic lesions | within 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Rex, Dr, Principal Investigator — University of Indiana Hospital; Douglas Morgan, Dr, Principal Investigator — University of North Carolina
Locations (4):
- United States (4):
  - University of Indiana Hospital, Indianapolis, Indiana
  - University of North Carolina, Chapel Hill, North Carolina
  - Digestive Care Inc., Beavercreek, Ohio
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia